CLINICAL TRIAL: NCT01190163
Title: Phase IV, Multicenter, Open Label, Randomized Trial to Compare the Effectiveness and Safety of the Dinoprostone Vaginal Pessary vs. Oxytocin for Women Requiring Cervical Ripening Prior to Induction of Labor
Brief Title: Open Label Comparative Trial of Dinoprostone Plus or Minus Oxytocin Versus Oxytocin Alone in Cervical Ripening for Labor Induction
Acronym: SOFTNES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was early terminated due to problems enrolling adequate number of patients
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE999901 CS01
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Vaginal Delivery; Cesarean Section
Keywords: Vaginal Birth delivery within 24 hours and C-section rate
MeSH Terms: interventions — Dinoprostone; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Dinoprostone
- B (Active Comparator)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Dinoprostone
  Arms: A
Drug: Oxytocin
  Arms: B

SUMMARY:
This is a comparative trial between oxytocin alone and dinoprostone for cervical ripening in unfavorable cervix pregnant women with 38 or more weeks of gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age ≥ 38 weeks
* Fetal cephalic presentation
* Bishop score < 6

Exclusion Criteria:

* No uterine scar (no previous delivery by caesarean section)
* No more than 3 previous vaginal births
* No condition that disallows use of prostaglandins for induction of labor
* Premature rupture of the membranes
* Oligohydramnios

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Vaginal birth delivery within 24 hours and C-section rate | 24 hours

SECONDARY OUTCOMES:
Treatment failure rate | 24 hours
Uterine hyperstimulation and/or fetal distress | 24 hours
Use of additional oxytocin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (4):
- Brazil (4):
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Hospital Municipal Universitário - Faculdade de Medicina do ABC, São Bernardo do Campo, São Paulo
  - Hospital M Boi Mirim, São Paulo, São Paulo
  - Hospital Maternidade Leonor Mendes de Barros, São Paulo, São Paulo